

Participant identification number

## **RECORD OF PARTICIPANT'S VERBAL CONSENT**

## **Understanding Patterns of Fatigue in Health and Disease**

The following is a telephone script and record of verbal consent for participants who indicate to the researchers that they would like to participate in the study. A copy of this consent form will be scanned or photocopied and sent to the participant via email or by post (according to their preference). Researcher introduces themself and the study and checks whether it is an appropriate time to conduct the consent process. Researcher checks participant's name and asks permission to audio-record the consent process. Audio-recorder is then turned on.

| Chief | Investigator: Dr Rosalind Adam | Researcher<br>initials |
|---|---|---|
| 1. | I confirm that I have read and understand the information sheet (version date) for the above study, have had the opportunity to ask questions, and have had these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. Only anonymised data collected up until the point of withdrawal may still be used in analysis. | |
| 3. | I agree to provide data collected via a wearable patch and a wrist worn device | |
| 4. | I agree to provide ratings of my fatigue via a smartphone app | |
| 5. | I agree to taking part in an interview with a researcher at the end of the study | |
| 6. | I agree to my interview being audio-recorded. I understand that my recording will be kept confidential and that anonymous quotations from recordings may be used in presentations | |
| | and publications. | Yes No |
| 7. | I agree to take part in a "feedback session" after my data have been analysed. I agree to this session being audio recorded. I understand that my recording will be kept confidential and that anonymous quotations from this session may be used in publications and presentation | |

IRAS Project ID: 317198



| Name of Researcher | Signature of Researcher | Date and Time | - |
|---|---|---|---|
| Name of Participant | | | |
| (If Participant agrees t | to participate, researcher asks the participant signs and dates below) | t to confirm their full name and | |
| 12. I agree to take p | part in the above study | | |
| related to this s | ne invited to take part in future ethically revientudy. I understand identifiable contact inforn<br>y and this information will be held in accorda | nation will be kept after the | Yes No |
| University of Ab | at data collected during the study may be loo<br>perdeen, the regulatory authorities or from N<br>his research. I give permission for these indivi | HS, where it is relevant to my | |
| findings are not | earchers can contact my general practitioner red during the study (for example, ECG chang or investigating, but that have been noted by ant) | es that the researchers were not | |
| College London, University of Gla information suc | data can be shared with the collaborating involversity of Cambridge, University of Lanca asgow and Panoramic Digital Health. I understh as contact details will only be shared when from one of these organisations to contact messession). | ester, Southampton University, stand that identifiable it is necessary for a research | |
| 8. I agree that Info | ormation about me can be stored on Universi<br>outer servers. | ty of | |

IRAS Project ID: 317198



IRAS Project ID: 317198